CLINICAL TRIAL: NCT00933023
Title: A Randomised Controlled Trial of Mild Versus Potent Topical Corticosteroids as Primary Treatment for Non-retractile Foreskin in Children.
Brief Title: Mild Versus Potent Corticosteroids as Treatment for Phimosis in Children
Acronym: TopSteP
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Patient numbers estimated to be too low to complete the trial in less than 10 years
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Anindya Niyogi, Clinical Research Fellow, Chelsea and Westminster NHS Foundation Trust
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TopSteP
Record Dates: First submitted 2009-07-06; First posted 2009-07-07 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Phimosis
MeSH Terms: conditions — Phimosis | interventions — Hydrocortisone; Betamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mild steroid (Experimental): 1%hydrocortisone for 8 weeks
  Interventions: Drug: hydrocortisone
- Potent Steroid (Experimental)
  Interventions: Drug: Betamethasone

INTERVENTIONS:
Drug: hydrocortisone — 1%hydrocortisone topical once daily for 8 weeks
  Arms: Mild steroid
Drug: Betamethasone — Betamethasone 0.1% topical once daily for 8weeks
  Arms: Potent Steroid

SUMMARY:
Topical steroids are used as treatment for non-retractile foreskin in children for decades, but, there are disagreement among physicians about the optimum potency of the agent used. This study is designed to determine any difference in the beneficial effects of mild versus potent topical corticosteroids in treatment of non-retractile foreskin in children.

ELIGIBILITY:
Inclusion Criteria:

* Children 2-16 with non-retractile foreskin

Exclusion Criteria:

* Balanitis xerotica obliterans, balanitis, <2yrs

Ages: 2 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Achievement of fully retractile foreskin with full exposure of glans at the end of therapy | 16 weeks

SECONDARY OUTCOMES:
Complications of topical corticosteroids | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anindya Niyogi, MBBS, MRCSEd, Principal Investigator — Research Fellow in Paediatric Surgery
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom